CLINICAL TRIAL: NCT00694044
Title: A Randomized, Investigator and Subject Blind, Sponsor Open Parallel Group Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pro-Cognitive Effects of Varenicline, Under Various Titration Schemes, in Healthy Elderly Non-Smoking Subjects
Brief Title: Evaluation of Varenicline Safety, Tolerability, Pharmacokinetics and Pro-Cognitive Effects in Healthy Elderly Non-Smoking Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: A3051106
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-06

CONDITIONS: Healthy; Non-Smoking
Keywords: Safety, Tolerability, Pharmacokinetics, Cognition
MeSH Terms: interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Weekly titration (Active Comparator)
  Interventions: Drug: varenicline
- Two Week QD (Active Comparator)
  Interventions: Drug: varenicline
- Two Week BID (Active Comparator)
  Interventions: Drug: varenicline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: varenicline — 0.5 mg once daily for 7days followed by 0.5 mg twice daily for 7days followed by 1mg twice daily for 7 days
  Other Names: Champix, Chantix
  Arms: Weekly titration
Drug: varenicline — 0.5 mg once daily for 14 days followed by 1 mg once daily for 7 days
  Other Names: Champix, Chantix
  Arms: Two Week QD
Drug: varenicline — 0.5 mg once daily for 14 days followed by 0.5 mg twice daily for 7 days
  Other Names: Champix, Chantix
  Arms: Two Week BID
Drug: Placebo — Placebo for 21 days
  Arms: Placebo

SUMMARY:
1. Characterize the tolerability and safety of repeated doses of varenicline in healthy non-smoking elderly subjects.
2. Describe the steady state pharmacokinetics of varenicline in healthy non-smoking elderly subjects.
3. Evaluate the potential effects of repeat doses of varenicline on cognition in healtly non-smoking elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy, Elderly (65-85 years inclusive), Non-smoker

Exclusion Criteria:

Creatinine Clearnace < 30 ml/min, Evidence or history of clinically significant, unstable diseases

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Tolerability and safety (adverse events, electrocardiogram, vital signs, clinical safety labs, self reported nausea visual analogue scales) | 21 days
Steady state pharmacokinetics | 21 days
Effects on cognition (computerized battery of cognitive tests) | 21 days

SECONDARY OUTCOMES:
No secondary outcomes. | Time frame n/a

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051106&StudyName=Evaluation%20of%20Varenicline%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20and%20Pro-cognitive%20Effects%20in%20Healthy%20Elderly%20Non-smoking%20Subjects